CLINICAL TRIAL: NCT04442555
Title: Treatment With the Ketone Body 3-hydroxybutyrate in Patients With Acute Heart Failure
Acronym: KETO-AHF1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kristian Hylleberg Christensen, MD, Principal Investigator, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KETO-AHF1 1-10-72-59-19
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-Hydroxybutyrate treatment (Experimental): HVMN Ketone Ester 0,5 g / kg
  Interventions: Dietary Supplement: HVMN Ketone Ester
- Placebo Treatment (Placebo Comparator): Maltodextrin-base isocaloric placebo
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: HVMN Ketone Ester — Commercially available ketone supplement
  Arms: 3-Hydroxybutyrate treatment
Dietary Supplement: Maltodextrin — Commercially available maltodextrin supplement
  Arms: Placebo Treatment

SUMMARY:
Background:

Acute heart failure is a potentially life-threatening condition, reaching mortality rates of up to 50% in advanced cases. The investigators have shown that infusion of ketone bodies increase cardiac output by 40% in stabile patients with chronic heart failure. However, there are no data showing the effects of ketone on patients with acute heart failure

Objectives:

To investigate the effect of ketone supplementation in patients with acute heart failure and cardiogenic shock, using two different types of oral ketone supplements.

Methods:

The investigators will conduct four randomized placebo-controlled studies, to investigate the hemodynamic effect of exogenous ketones in acute heart failure and cardiogenic shock.

Perspectives:

The present study will determine the potential beneficial effects of ketone supplements in patients with acute heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with worsening HF or de novo diagnosis of HF
* LVEF < 50%
* Treatment with intravenous loop diuretics during the hospitalization and/or increased dosage of oral diuretics.

Exclusion Criteria:

* Cardiogenic shock
* Systolic Blood Pressure <85 mmHg
* Acute myocardial infarction other than type II <5 days prior to randomization *
* Severe uncorrected cardiac valve disease
* Expected or possible need for hemodialysis as judged by the investigator
* Ongoing inotropic treatment
* Possible need for advanced heart failure treatment (LVAD, heart transplantation) as judged by the investigator.
* Ongoing, severe infection
* Severe respiratory distress (SAT<90% or RF> 24/min or receiving more than 2 l O2/min or intubated)
* Atrial Fibrillation with heart >120 beats per minute
* Inability to cooperate to or accept oral intake of food, including presence of major gastrointestinal discomfort.

  * If suspected or confirmed acute myocardial infarction as cause of acute heart failure, patients can be recruited 5 days after hospitalization in the absence of malignant arrhythmias (e.g. ventricular tachycardia) or clinically significant residual angina pectoris.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac Output (L/min) | 3 hours - Area under the curve
  Right Heart Catherization
Left Ventricular Ejection Fraction | 3 hours - Area under the curve
  Echocardiography

SECONDARY OUTCOMES:
Left Ventricular Outflow Tract Velocity Time Integral (cm) | 3 hours - Area under the curve
  Echocardiography
Left Ventricular Filling Pressure (mmHg) | 3 hours - Area under the curve
  Right Heart Catherization

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No